CLINICAL TRIAL: NCT03169543
Title: Neural Mechanisms Underlying the Antidepressant Effects of Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 811678
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep deprivation (Experimental): 36-hours of total sleep deprivation
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — 36-hours total sleep deprivation

SUMMARY:
From 40 to 60% of patients with depression experience a rapid and significant improvement of mood with one night of sleep deprivation (SD). The neural mechanisms underlying this effect have not been elucidated. Recent advances in functional neuroimaging have provided new opportunities to investigate state changes in regional brain function, along with a better understanding of the neural networks affected by depression and SD. Here we propose to study a group of N=48 antidepressant-free male and female patients with current depression symptom and N=12 healthy controls with no history of mood disorders before and after SD to provide mechanistic insight into the neural substrates underlying the antidepressant effects of SD. We hypothesize that SD-induced concurrent functional activity and connectivity changes in multiple brain networks related to different depressive symptom dimensions including emotion regulation, attention, arousal, self-referential, and reward processing will underlie the rapid and transient antidepressant effects of SD. Using an ABA design, multimodal brain imaging along with more traditional electroencephalographic (EEG) and neurobehavioral testing data will be acquired at baseline after normal sleep, during one night of total SD, and after one night of recovery sleep using a 5-day in laboratory protocol during which subjects will be continuously monitored by trained staff.

ELIGIBILITY:
Inclusion Criteria:

* Current depression as assessed on the HDRS-17 (for depressed group only)
* Body mass index within 15% of normal
* Stable, normally-timed sleep-wake cycle defined by: a. Habitual nocturnal sleep duration between 6h and 9h. b. Habitual morning awakening between 0600h and 0800h.
* Able to comprehend English, as all questionnaires are in this language
* Ability to provide informed consent

Exclusion Criteria:

* Shift work, transmeridian travel or irregular sleep/wake routine in past 60 days
* A sleep disorder other than insomnia
* History of bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia and other psychotic disorders
* No history of depression for the control group.
* Alcohol or drug abuse in the past year
* A current smoker.
* Any acute or chronic, debilitating medical conditions, epilepsy, or thyroid disease.
* Metallic implants, pacemakers or tattoos, or history of working in metal workshops.
* Claustrophobic, or intolerant of the scanner environment.
* For women, pregnancy will exclude participation.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in HAMD-NOW scores | Each morning for 4 days
  Total score on a modified Hamilton Depression Inventory that assesses mood symptoms in the moment.

SECONDARY OUTCOMES:
Change in neuroimaging | Each morning for 3 days
  Resting-state brain functional connectivity on fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gehrman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No